CLINICAL TRIAL: NCT03128983
Title: Variations of Physiological Data Throughout the Menstrual Cycle
Brief Title: Physiological Data in the Menstrual Cycle
Acronym: PDMC
Status: Completed | Type: Observational
Sponsor: Ava AG (Industry)
Collaborators: University Hospital, Zürich (Other); Centre Suisse d'Electronique et de Microtechnique (CSEM), Switzerland (Unknown); Empa, Swiss Federal Laboratories for Materials Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: Emilia
Record Dates: First submitted 2017-04-21; First posted 2017-04-25 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Fertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Participants wear a sensor bracelet for collecting physiological data and conducted urine tests to estimate the day of ovulation

SUMMARY:
Research results suggest changes of physiological parameters such as heart rate, respiration, skin conductance response, sleep duration, sleep quality and skin perfusion during the menstrual cycle. Latest fitness trackers allow to conveniently and non-invasively record these parameters. The present study aims to evaluate whether there is a correlation between physiological parameters and the menstrual cycle i.e. ovulation as measured by a urine ovulation test and the onset of menses. To collect data women will wear two smartwatches and a smartshirt at night. All three devices are CE-approved for sports and fitness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-pregnant women aged 20-40 years (healthy volunteers)
* Regular cycling (28 days +/- 2)
* Non-hormonal contraception methods used
* German-speaking
* Written informed consent to participate in the study

Exclusion Criteria:

* Any health-related issues that may affect menstrual cycle
* Any consumption of medication or other substances that may affect the menstrual cycle or any of the physiological parameters investigated
* Frequent travel between time zones
* Sleeping disorders

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The monitoring of menstrual cycles requires female participants.
Study Population: A maximum of 50 healthy, 20-40 years old, non-pregnant women will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between menstrual cycle dynamics and physiology | During 1 menstrual cycle between 24 days and 35 days
  Correlation between a combination of the physiological parameters heart rate, respiration, skin conductance response, sleep duration, sleep quality and skin perfusion and menstrual cycle dynamics.

IPD SHARING:
Plan to Share IPD: No